CLINICAL TRIAL: NCT04731324
Title: A Phase 1, Prospective Open Label, Single Dose, Single Arm Study of ZYIL1 Administered Via Oral Route to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Healthy Adult Human Subjects
Brief Title: Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of ZYIL1 Following Oral Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYIL1 1001; CTRI/2020/12/030045 (Registry Identifier: Clinical Trial Registry of India)
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: COVID 19; NLRP3; NLPR3 Inflammasone inhibitor
MeSH Terms: conditions — COVID-19 | interventions — ZYIL1

STUDY DESIGN:
Intervention Model Description: A phase 1, prospective open label, single dose, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZYIL1 Capsule (Experimental): six subjects will be recruited in each cohort. safety data up to day 3 will be evaluated to determine whether progression to the subsequent dose Cohort is indicated. Single dose will be administered in ascending manner starting from 25 mg.
  Interventions: Drug: ZYIL1 capsule

INTERVENTIONS:
Drug: ZYIL1 capsule — NLRP3 inflammasome inhibitor

SUMMARY:
ZYIL1 is a novel oral selective NLRP3 inflammasome inhibitor which prevents NLRP3-induced ASC oligomerization, thus inhibiting NLRP3 inflammasome pathway. ZYIL1 is expected to show benefit in patients demonstrating cytokine, like IL1β flare, including those exhibiting cytokine storm related to COVID-19 and other viral inflammatory diseases.

DETAILED DESCRIPTION:
It is an open label, study designed to evaluate safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) following a single-oral dose administration of ZYIL1 to healthy subjects aged between 18-55 years old (Both Inclusive).

It will be conducted in up to 7 cohorts of 6 subjects each. Each cohort will be enrolled within a 28 day screening period to ensure subjects meet all the inclusion criteria and none of the exclusion criteria. Subjects will be administered single oral dose of ZYIL1 on Day 1.

In this study each cohort containing six subjects will be given a single oral dose of ZYIL1 in ascending manner. Initially, up to 3 cohorts of 18 subjects will be enrolled and dosed. Interim analysis will be done after completion of three cohorts and submitted to Central Licensing Authority of India(CLA). Further cohorts (i.e. cohort S4 onwards) will be conducted after obtaining approval of CLA.

This is the first administration of ZYIL1 in humans; therefore, study design adjustments may be made based on emerging data from each dose cohort based on review of preliminary safety, tolerability, and PK results.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-lactating non-pregnant female between 18 and 55 years of age at the time of signing the informed consent form (ICF). (Both inclusive).
2. Body mass index of 18.5 to 30.0 kg/m2 (Both inclusive) with a body weight of 50 to 100 kg (Both inclusive).
3. Normal QTc interval at screening and Check In [QTcF ≤450 ms]
4. Male subjects must agree to use adequate contraception methods during the study and be willing and able to continue contraception for 90 days after administration of study treatment.
5. Capable of giving written informed consent, which includes compliance with the study procedures, restrictions, and requirements listed in the protocol.
6. Subjects who, in the opinion of the Investigator, are healthy as determined by their pre study medical history, clinical examination, 12-lead ECG and clinical laboratory tests within the institutional normal range or judged as not clinically significant by the Investigator, including the following parameters: hematology, serum biochemistry, urinalysis, and serology
7. Female subjects with history of sterility or at least 1 year menopause or use of long acting non hormonal contraceptive measures (e.g., intrauterine device) and be willing and able to continue contraception for 90 days after administration of study treatment.

Exclusion Criteria:

1. History or presence of alcoholism or drug abuse within the past 1 year.
2. Presence or history of any of the following disorders/disease within the past 3 months, that might have impact on the clinical trial as per the investigator discretion: cardiovascular, cerebrovascular, dermatological, gastrointestinal, gynecological, hematological, hepatic, malignancy, metabolic, musculoskeletal, neurological, urological, psychiatric, renal, respiratory, venereal, any other major disorders
3. History of clinically significant hypersensitivity, intolerance, or allergies, as determined by the Investigator.
4. History of COVID-19 infection within 14 days or contact with a confirmed active COVID-19 positive patient within 14 days; or positive COVID-19 test within 5 days of Check-in. .
5. History or presence of smoking or consumption of tobacco/nicotine products within the past 1 year.
6. Difficulty with donating blood.
7. Systolic blood pressure more than 140 mmHg or less than 100 mmHg or diastolic blood pressure more than 90 mmHg or less than 60 mmHg.
8. Pulse rate less than 55/minute or more than 100/minute.
9. Any clinically significant laboratory or ECG findings during screening
10. Surgery within last 3 months or planned major surgery within next 3 months from the date of screening (other than minor cosmetic surgery and minor dental surgery).
11. Subjects who have recent illness (eg, fever) within 14 days of check-in
12. Volunteers who have participated in any drug research study within past 3 months.
13. Volunteers who have donated one unit (350 ml) of blood in the past 3 months.
14. Has used prescription drugs and other substances (eg, dietary or herbal supplements such as St John's Wort) known to be either significant enzyme inducers or enzyme inhibitors within 4 weeks of Day 1, or use of grapefruit or similar substances (Seville oranges or marmalade, grapefruit juice, grapefruit hybrids, pomelos, exotic citrus fruits or fruit juices) within 7 days of Day 1.
15. Use of any over-the-counter (OTC), any prescription medications or alternative tradition of medicine (herbal medicines, homoeopathy, Siddha, Unani, etc.) within the 15 days or 5 half-lives (whichever is longer), prior to receiving study drug that might have impact on the clinical trial as per the investigator discretion.
16. A positive urine drugs of abuse test or positive alcohol test at check-in.
17. History of, or positive screening test for, hepatitis C infection (defined as positive for hepatitis C virus antibody), hepatitis B infection (defined as positive for hepatitis B surface antigen), or human immunodeficiency virus I or II.
18. Any disorder that, in the Investigator's opinion, may interfere with study compliance, such as significant mental, nervous disorder or other illness. In making this assessment, the Investigator must refer to the study information provided including the Investigator's Brochure.
19. Inability to be venipunctured or tolerate venous puncture.
20. Any condition or abnormal baseline findings that in the Investigator's judgment might increase the risk to the subject or decrease the chance of obtaining satisfactory data needed to obtain the objective of the study.
21. Other unspecified reasons that, in the opinion of the Investigator or the Sponsor, make the subject unsuitable for the study.
22. Female subjects who are pregnant, currently breastfeeding, or attempting to conceive.

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse event of ZYIL1 following a single oral dose in healthy subjects | Baseline to Day 3
  The Common Terminology Criteria for Adverse Event (CTCAE) (Version 5.0 or higher) system will be used for reporting and grading

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Predose; 0.5 hour; 1 hour; 1.5 hour; 2 hour; 3 hour; 4 hour; 5 hour, 6 hour; 8 hour; 12 hour, 24 hour and 48 hour
  At each dose level, blood samples will be withdrawn for the evaluation of pharmacokinetic.

OTHER OUTCOMES:
Time to reach maximum plasma concentration (Tmax) | Predose; 0.5 hour; 1 hour; 1.5 hour; 2 hour; 3 hour; 4 hour; 5 hour, 6 hour; 8 hour; 12 hour, 24 hour and 48 hour
  At each dose level, blood samples will be withdrawn for the evaluation of pharmacokinetic.
Area under the curve from the time of dosing to the last measurable concentration (AUC0-t) | Predose; 0.5 hour; 1 hour; 1.5 hour; 2 hour; 3 hour; 4 hour; 5 hour, 6 hour; 8 hour; 12 hour, 24 hour and 48 hour
  At each dose level, blood samples will be withdrawn for the evaluation of pharmacokinetic.
Terminal half life (t1/2) | Predose; 0.5 hour; 1 hour; 1.5 hour; 2 hour; 3 hour; 4 hour; 5 hour, 6 hour; 8 hour; 12 hour, 24 hour and 48 hour
  At each dose level, blood samples will be withdrawn for the evaluation of pharmacokinetic.
Elimination rate constant (λz) | Predose; 0.5 hour; 1 hour; 1.5 hour; 2 hour; 3 hour; 4 hour; 5 hour, 6 hour; 8 hour; 12 hour, 24 hour and 48 hour
  At each dose level, blood samples will be withdrawn for the evaluation of pharmacokinetic.
Clearance (CL/F) | Predose; 0.5 hour; 1 hour; 1.5 hour; 2 hour; 3 hour; 4 hour; 5 hour, 6 hour; 8 hour; 12 hour, 24 hour and 48 hour
  At each dose level, blood samples will be withdrawn for the evaluation of pharmacokinetic.
Volume of distribution (Vd) | Predose; 0.5 hour; 1 hour; 1.5 hour; 2 hour; 3 hour; 4 hour; 5 hour, 6 hour; 8 hour; 12 hour, 24 hour and 48 hour
  At each dose level, blood samples will be withdrawn for the evaluation of pharmacokinetic.
Amount recovered in Urine | Pre dose, 0-4 hours, 4-8 hours, 8-12 hours , 12-24 hours, 24-36 hours and 36 - 48 hours
  Urine will be collected following IMP administrations on Day 1.The quantity of total urine collected at each time point will be recorded for calculating total urine output up to 48 hours.
Percent recovered in urine | Pre dose, 0-4 hours, 4-8 hours, 8-12 hours , 12-24 hours, 24-36 hours and 36 - 48 hours
  Urine will be collected following IMP administrations on Day 1.The quantity of total urine collected at each time point will be recorded for calculating total urine output up to 48 hours.
Levels of IL-1β based on ex vivo LPS/ATP stimulation assay | Pre-dose, 3 hour, 6 hour, 12 hour and 24 hour
  At each dose level, blood samples will be withdrawn for the evaluation of pharmacodynamics
Levels of IL-18 based on ex vivo LPS/ATP stimulation assay | Pre-dose, 3 hour, 6 hour, 12 hour and 24 hour
  At each dose level, blood samples will be withdrawn for the evaluation of pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Dr Deven Parmar, MD, Study Chair — Cadila Healthcare Ltd.
Locations (1):
- Zydus Research Centre, Ahmedabad, Gujarat, India

REFERENCES:
- [Derived] Parmar DV, Kansagra KA, Momin T, Patel HB, Jansari GA, Bhavsar J, Shah C, Patel JM, Ghoghari A, Barot A, Sharma B, Viswanathan K, Patel HV, Jain MR. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Oral NLRP3 Inflammasome Inhibitor ZYIL1: First-in-Human Phase 1 Studies (Single Ascending Dose and Multiple Ascending Dose). Clin Pharmacol Drug Dev. 2023 Feb;12(2):202-211. doi: 10.1002/cpdd.1162. Epub 2022 Sep 5. PMID 36065092